CLINICAL TRIAL: NCT01502228
Title: PET/CT Assessment of Tumor Perfusion in Patients With Renal Cell Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No further funding
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Theodore Logan, Associate Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IUCRO-0279
Record Dates: First submitted 2011-12-28; First posted 2011-12-30 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Magnetic Resonance Spectroscopy; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 62Cu-ETS PET assessment (Experimental): CT scan for attenuation correction; 15O-water administered by intravenous injection and 6-minute dynamic PET imaging; 62Cu-ETS administered by intravenous injection; Dynamic PET acquisition for 6-minutes; Whole-body PET acquisition from 6-20 minutes post-62Cu-ETS injection
  Interventions: Drug: 150-Water; Drug: 62Cu-ethylglyoxal bis; Procedure: Positron Emission Tomography; Drug: Sunitinib

INTERVENTIONS:
Drug: 150-Water — Patients will be imaged immediately before, and between 14-28 days after initiation of Sunitinib therapy, in the single bed position using the Siemens Biograph 64 TruePoint system located in the clinical facilities of the I.U. Cancer Center. Administer 15O-water at 50 mCi/dose, IV.
Drug: 62Cu-ethylglyoxal bis — Imaging with 62Cu-ETS will be done immediately following imaging with 150-water. Patients will be imaged immediately before, and between 14-28 days after, initiation of Sunitinib therapy using the Siemens Biograph 64 TruePoint system located in the clinical facilities of the I.U. Cancer Center. Administer 62Cu-ETS in the range of 20-25 mCi/Dose, IV.
Procedure: Positron Emission Tomography — PET Scan
  Other Names: Seimens Biograph 64 TruePoint system
Drug: Sunitinib

SUMMARY:
Given the growing importance of anti-angiogenic therapies in the treatment of metastatic renal carcinoma, it is expected that this trial will establish the preliminary data needed to apply for funding of a larger clinical investigation of the potential role of PET perfusion imaging in management of renal carcinoma, and potentially other cancers.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a witnessed, informed consent and authorization for the release of health information.
* Patients with a diagnosis of relapsed Stage IV renal cell cancer that are medically unresponsive to prior treatment or surgically unresectable and with metastases that fall within the PET/CT field-of-view that can include the heart.
* Being considered for systemic therapy with Sunitinib

Exclusion Criteria:

* Women who are pregnant, breast-feeding, or of childbearing potential and not using birth control
* Having no telephone or a reliable way in which study personal can contact them
* Subjects who are claustrophobic and cannot tolerate imaging procedures
* Subjects who weigh > 350 lb. (upper weight limit of scanner beds)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Fletcher, M.D., Principal Investigator — Indiana University, Radiology; Theodore Logan, M.D., Principal Investigator — Indiana University, Dept. Medicine (Hem/Onc)
Locations (1):
- Indiana University Simon Cancer Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 09008-12(1011004283)-PT/CT Assessment of Tumor Perfusion in Patients with RCC — https://www.indianactsi.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol has 14 patients. Originally, 15 patients were planned, but lack of funding did not allow the final patient to be enrolled.
Groups:
- 62Cu-ETS PET Assessment: CT scan for attenuation correction; 15O-water administered by intravenous injection and 6-minute dynamic PET imaging; 62Cu-ETS administered by intravenous injection; Dynamic PET acquisition for 6-minutes; Whole-body PET acquisition from 6-20 minutes post-62Cu-ETS injection 150-Water: Patients will be imaged immediately before, and between 14-28 days after initiation of Sunitinib therapy, in the single bed position using the Siemens Biograph 64 TruePoint system located in the clinical facilities of the I.U. Cancer Center. Administer 15O-water at 50 mCi/dose, IV.
  62Cu-ethylglyoxal bis: Imaging with 62Cu-ETS will be done immediately following imaging with 150-water. Patients will be imaged immediately before, and between 14-28 days after, initiation of Sunitinib therapy using the Siemens Biograph 64 TruePoint system located in the clinical facilities of the I.U. Cancer Center. Administer 62Cu-ETS in the range of 20-25 mCi/Dose, IV. Positron Emission Tomography: PET Scan Sunitinib
Period: Overall Study
Arm/Group | 62Cu-ETS PET Assessment
Started | 14
Completed | 13
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | 62Cu-ETS PET Assessment
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Where 62Cu-ETS PET and 15O-water PET Was Obtained
Description: Number of patients who had at least a baseline measurement of 62Cu-ETS PET and 15O-water PET
Time Frame: Baseline
Population: All Patients Enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | 62Cu-ETS PET Assessment
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Maximum Standard Uptake Value (SUV) for Lesion Data
Description: Average values of the magnitude of tumor perfusion before and 14-28 days after initiation of Sunitinib treatment as measured by the maximum standard uptake value for all the lesion data. Standard uptake values were calculated as the ratio of the image derived radioactivity concentration and the whole body concentration of the injected radioactivity tracer. There were 14 patients who had a baseline reading and 12 patients who had a reading after treatment.
Time Frame: Baseline and 14-28 days after initiation of Sunitinib
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | 62Cu-ETS PET Assessment
Number analyzed (Participants) | 14
SUV
  Baseline | 5.84 (2.03)
  After Treatment | 4.86 (2.50)

ADVERSE EVENTS:
Time Frame: up to 3 years
Arm/Group | 62Cu-ETS PET Assessment
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 11/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 62Cu-ETS PET Assessment (N=14)
Anemia (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Fever (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Dysgeusia (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 3
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes